CLINICAL TRIAL: NCT00440557
Title: A Randomized, Open Label, Multicenter Study of Epoetin Alfa Comparing Two Extended-Dosing Regimens, Once-Weekly and Every-Two-Weeks, With the Three-Times-Weekly Dosing Regimen for Initiation and Maintenance Treatment in Anemic Subjects With Chronic Kidney Disease
Brief Title: An Efficacy and Safety Study of Epoetin Alfa for Initiation and Maintenance Treatment of Patients With Anemia Associated With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR010411; EPOAKD3001 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Anemia
Keywords: Anemia; Chronic Kidney disease; Kidney disease; Epoetin alfa; Procrit
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Diseases | interventions — Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TIW: Epoetin alfa 3 injections Weekly/Once Weekly (Experimental): Participants will be administered with epoetin alfa 3 times weekly for 22 weeks (initial subcutaneous (SC) dose 50 IU/kg), then once weekly, for 22 weeks (initial SC dose 10,000 IU)
  Interventions: Drug: Epoetin alfa 3 times weekly /once weekly
- QW: Epoetin alfa once weekly (Experimental): Participants will be administered with epoetin alfa once weekly for 44 weeks (initial subcutaneous dose 10,000 IU).
  Interventions: Drug: Epoetin alfa once weekly
- Q2W: Epoetin alfa once every two weeks (Experimental): Participants will be administered with epoetin alfa once every 2 weeks for 44 weeks (initial subcutaneous dose 20,000 IU).
  Interventions: Drug: Epoetin alfa once every two weeks

INTERVENTIONS:
Drug: Epoetin alfa 3 times weekly /once weekly — Epoetin alfa will be administered as a SC injections at initial dose of 50 IU/kg (3 times weekly for 22 weeks) and at initial dose of 10000 IU (once weekly for 22 weeks)
  Other Names: PROCRIT
  Arms: TIW: Epoetin alfa 3 injections Weekly/Once Weekly
Drug: Epoetin alfa once weekly — Epoetin alfa will be administered as a SC injection at initial dose of 10000 IU (once weekly for 44 weeks).
  Other Names: PROCRIT
  Arms: QW: Epoetin alfa once weekly
Drug: Epoetin alfa once every two weeks — Epoetin alfa will be administered as a SC injection at initial dose of 20000 IU (once every 2 weeks for 44 weeks).
  Other Names: PROCRIT
  Arms: Q2W: Epoetin alfa once every two weeks

SUMMARY:
The purpose of this study is to demonstrate that once weekly and once every-2-weeks treatment with epoetin alfa, in patients with anemia associated with chronic kidney disease, is not less effective than the approved treatment with epoetin alfa that is given 3 times weekly with respect to changes in hemoglobin.

DETAILED DESCRIPTION:
This is a open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), multicenter study designed to show that 2 alternative dosing regimens, once weekly and once every-2-weeks (given at doses equivalent to 50 IU/kg 3 times a week) are not inferior to the 3-times-weekly dosing regimen. Approximately 375 patients with anemia will be enrolled in this study. Patients will be randomly assigned to receive epoetin alfa by subcutaneous (SC) injection according to one of the following 3 regimens: 3 times weekly (Group 1), once weekly (Group 2), or once every 2 weeks (Group 3) for 22 weeks. Thereafter, patients in Group 1 will be switched to the once-weekly dosing regimen for an additional 22 weeks, and patients in Groups 2 and 3 will continue their current treatment for an additional 22 weeks. The total duration of the open-label treatment phase is 44 weeks which will include initiation and maintenance treatment periods (with the goal of increasing, then maintaining, the hemoglobin level between 11.0 and 11.9 g/dL inclusive) and a safety period (to assess longer exposure to epoetin alfa treatment and any period of hemoglobin instability during the transition from 3-times-weekly to once-weekly dosing). Starting doses of epoetin alfa in the 3-times-weekly, once-weekly, and every-2-weeks groups will be 50 IU/kg, 10,000 IU, and 20,000 IU, respectively; thereafter adjusted according to weekly hemoglobin concentrations. Safety evaluations will include assessment of adverse events, laboratory tests, physical examinations, and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for chronic kidney disease, defined as a glomerular filtration rate (GFR) more than or equal to 15 mL/min per 1.73 m2 and less than 60 mL/min per 1.73 m2 (Stages 3 and 4) as calculated by the central laboratory
* Require support of an erythropoietin receptor agonist

Exclusion Criteria:

* Uncontrolled hypertension
* Serum ferritin level less than 50 ng/mL
* Serum iron overload
* Severe congestive heart failure
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (62):
- United States (61):
  - Glendale, Arizona
  - Tempe, Arizona
  - Chula Vista, California
  - Long Beach, California
  - Los Angeles, California
  - Lynwood, California
  - Riverside, California
  - San Diego, California
  - Visalia, California
  - Whittier, California
  - Yuba City, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Thornton, Colorado
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Orlando, Florida
  - Palm Beach Gardens, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Carrollton, Georgia
  - Macon, Georgia
  - Statesboro, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Methuen, Massachusetts
  - Plymouth, Massachusetts
  - Flint, Michigan
  - Hackensack, New Jersey
  - Old Bridge, New Jersey
  - Vineland, New Jersey
  - Albuquerque, New Mexico
  - Great Neck, New York
  - New Hartford, New York
  - New York, New York
  - Springfield Gardens, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Maumee, Ohio
  - Doylestown, Pennsylvania
  - Easton, Pennsylvania
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Wynnewood, Pennsylvania
  - Bamberg, South Carolina
  - Orangeburg, South Carolina
  - Sumter, South Carolina
  - Dyersburg, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Chesapeake, Virginia
  - Fairfax, Virginia
  - Hampton, Virginia
  - Richmond, Virginia
  - Tacoma, Washington
- Caguas, Puerto Rico

REFERENCES:
- [Derived] Pergola PE, Gartenberg G, Fu M, Wolfson M, Rao S, Bowers P. A randomized controlled study of weekly and biweekly dosing of epoetin alfa in CKD Patients with anemia. Clin J Am Soc Nephrol. 2009 Nov;4(11):1731-40. doi: 10.2215/CJN.03470509. Epub 2009 Sep 17. PMID 19808215
- See also: A Randomized,Open-Label, Multicenter Study of Epoetin Alfa Comparing Two Extended-Dosing Regimens,OnceWeekly and EveryTwoWeeks,With the ThreeTimesWeekly Dosing Regimen for Initiation & Maintenance Treatment in Anemic Subjects With Chronic Kidney Disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=32&filename=CR010411_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated 29 August 2006 and completed on 21 February 2008. Subjects were screened for eligibility at 64 investigative sites within the U.S. Three hundred seventy-five subjects (intent to treat) were randomly assigned to a treatment group by 52 investigators from 56 sites. Safety population consisted of 373 subjects.
Groups:
- Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW): Epoetin alfa 3 times weekly for 22 weeks (initial subcutaneous (SC) dose 50 IU/kg), then once weekly, for 22 weeks (initial SC dose 10,000 IU)
- Epoetin Alfa:Once Weekly (QW): Epoetin alfa once weekly for 44 weeks (initial subcutaneous dose 10,000 IU)
- Epoetin Alfa:Once Every Two Weeks (Q2W): Epoetin alfa once every 2 weeks for 44 weeks (initial subcutaneous dose 20,000 IU)
Period: Overall Study
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Started | 123 (Safety population defined as all subjects who received at least 1 injection of study drug.) | 125 (Safety population defined as all subjects who received at least 1 injection of study drug.) | 125 (Safety population defined as all subjects who received at least 1 injection of study drug.)
Completed | 98 | 96 | 90
Not Completed | 25 | 29 | 35
Not completed — Withdrawal by Subject | 10 | 5 | 11
Not completed — Lost to Follow-up | 1 | 2 | 6
Not completed — Adverse Event | 3 | 3 | 5
Not completed — Death | 2 | 6 | 3
Not completed — Began Dialysis | 4 | 1 | 4
Not completed — Principal Investigator decision | 0 | 3 | 1
Not completed — Patient moved | 1 | 2 | 1
Not completed — Principal Investigator's office closed | 3 | 6 | 4
Not completed — Patient transferred to nursing home | 0 | 1 | 0
Not completed — Patient had surgery | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W) | Total
Number analyzed (Participants) | 123 | 125 | 125 | 373
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 43 | 44 | 120
  >=65 years | 90 | 82 | 81 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (13.02) | 68.9 (11.86) | 68.9 (13.02) | 69.6 (12.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 80 | 85 | 242
  Male | 46 | 45 | 40 | 131

OUTCOME MEASURES:

1. Primary Outcome: Change in Hb Concentration (g/dL) From Baseline to the Average of the Last 8 Weeks of Treatment Through Week 22
Description: The change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included in calculating the average Hb during the last 8 weeks of treatment through Week 22.
Time Frame: From baseline through Week 22
Population: Modified Intent-To-Treat (mITT) population. The mITT population was defined as all participants who were randomized and had at least 1 postrandomization hemoglobin concentration measurement.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 121 | 124 | 123
g/dL | 1.81 (0.910) | 1.59 (0.997) | 1.27 (0.906)
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); The null hypothesis is the mean change in Hb concentration from baseline to the average of the last 8 weeks of treatment (tX) through Week 22 in the QW group is not lower than that of the TIW group by more than 1 g/dL; Test type: Non-Inferiority or Equivalence — Assuming a difference in the mean change in Hb from baseline to the average of the last 8 weeks of treatment through Week 22 of -0.3 g/dL between standard-tx group (TIW) and test-tx group (QW), a pooled standard deviation of 1.7 g/dL, and a noninferiority margin of 1 g/dL, a sample size of approximately 250 participants (125 per group) will provide 90% power to demonstrate that the test treatment group is not inferior to the standard-treatment group for an overall 2-sided 0.05 significance level; This comparison between QW and TIW was performed prior to comparing Q2W with TIW in the statistical analysis 2 according to a planned stepdown procedure for controlling multiplicity; Difference of Least Squares Means = -0.17, 95% CI [-0.380 to 0.037], Standard Error of Mean 0.106
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); The null hypothesis is the mean change in Hb concentration from baseline to the average of the last 8 weeks of treatment through Week 22 in the Q2W group is not lower than that of the TIW group by more than 1 g/dL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Since the non-inferiority was declared in the statistical analysis 1, this comparison between Q2W and TIW was then performed according to a planned stepdown procedure for controlling multiplicity; Difference of Least Squares Means = -0.43, 95% CI [-0.641 to -0.221], Standard Error of Mean 0.107

2. Other Pre Specified Outcome: Participants Who Exceeded a Hb Concentration of 11.9 g/dL During First 22 Weeks of Treatment
Description: The change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. participants who exceed a Hb value of 11.9 g/dL at least once were included in the numerator of the percentage calculation.
Time Frame: From baseline to Week 22
Population: Safety population. The safety population was defined as all participants who received at least 1 injection of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 123 | 125 | 125
participants | 106 | 98 | 89
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; Difference in Percentage of Participants = -7.8, 95% CI [-17.2 to 1.7]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; Difference in Percentage of Participants = -15.0, 95% CI [-25.0 to -5.0]

3. Other Pre Specified Outcome: Maximum Hb Concentration (g/dL) During First 22 Weeks of Treatment
Description: The change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. A maximum Hb observation was identified for each participant during the first 22 weeks of treatment.
Time Frame: From baseline to Week 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 123 | 125 | 125
g/dL | 12.87 (1.176) | 12.61 (1.158) [-0.564 to 0.043] | 12.42 (1.310) [-0.755 to -0.147]
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; ANOVA; Difference of Least Squares Means = -0.26, 95% CI [-0.564 to 0.043]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; ANOVA; Difference of Least Squares Means = -0.45, 95% CI [-0.755 to -0.147]

4. Other Pre Specified Outcome: Participants Who Met or Exceeded Hb Rate of Rise >=1.0 g/dL/2 Weeks During First 22 Weeks of Treatment
Description: Change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. Participants who met or exceeded a Hb Rate of Rise (RR) of 1.0 g/dL/2 weeks at least once were included in the numerator of the percentage calculation.
Time Frame: From baseline to Week 22
Population: Safety population. The safety population was defined as all subjects who received at least 1 injection of study drug.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 123 | 125 | 125
participants | 119 | 116 | 114
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; Difference in Percentage of Participants = -3.9, 95% CI [-9.5 to 1.6]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; Difference in Percentage of Participants = -5.5, 95% CI [-11.4 to 0.3]

5. Other Pre Specified Outcome: Participants Who Met or Exceeded Hb Rate of Rise >=1.5 g/dL/2 Weeks During First 22 Weeks of Treatment
Description: Change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. Participants who met or exceeded a Hb Rate of Rise (RR) of 1.5 g/dL/2 weeks at least once were included in the numerator of the percentage calculation.
Time Frame: From baseline to Week 22
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 123 | 125 | 125
participants | 87 | 85 | 76
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; Difference in Percentage of Participants = -2.7, 95% CI [-14.2 to 8.7]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; Difference in Percentage of Participants = -9.9, 95% CI [-21.7 to 1.8]

6. Other Pre Specified Outcome: Particpants Who Met or Exceeded Hb Rate of Rise >=2.0 g/dL/2 Weeks During First 22 Weeks of Treatment
Description: Change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. Participants who met or exceeded a Hb Rate of Rise (RR) of 2.0 g/dL/2 weeks at least once were included in the numerator of the percentage calculation.
Time Frame: From baseline to Week 22
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 123 | 125 | 125
participants | 47 | 51 | 44
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; Difference in Percentage of Participants = 2.6, 95% CI [-9.6 to 14.8]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; Difference in Percentage of Participants = -3.0, 95% CI [-15.0 to 9.0]

7. Post Hoc Outcome: Maximum (Max) Hb Rate (g/dL/2 Weeks) of Rise During First 22 Weeks of Treatment
Description: Change is calculated as mean hemoglobin (Hb) over last 8 wks subtracts baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. Max Hb RR observation was identified for each participant during the 1st 22 wks of treatment. This was the max RR in hemoglobin over any 2-wk period per participant.
Time Frame: From baseline to Week 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: g/dL/2 weeks
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 123 | 125 | 125
g/dL/2 weeks | 1.99 (0.839) | 2.02 (1.008) [-0.210 to 0.270] | 1.92 (1.027) [-0.315 to 0.166]
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; ANOVA; Difference of Least Squares Means = 0.03, 95% CI [-0.210 to 0.270]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; ANOVA; Difference of Least Squares Means = -0.07, 95% CI [-0.315 to 0.166]

8. Secondary Outcome: Participants With an Increase of ≥1 g/dL in Hb Concentration From Baseline by Week 9
Description: The change is calculated as average hemoglobin (Hb) over the last 8 weeks subtracts the baseline Hb. Only Hb measurements up until a participant receives a transfusion or begins dialysis were included. Hb increase is defined as the post-baseline Hb level minus the baseline Hb level.
Time Frame: From baseline to Week 9
Population: Modified Intent-To-Treat (mITT) population. The mITT population was defined as all participants who were randomized and had at least 1 postrandomization Hb concentration measurement.
Measure: Number; unit: participants
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Number analyzed (Participants) | 121 | 124 | 124
participants | 116 | 108 | 106
Statistical Analysis 1: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Weekly (QW); Test type: Superiority or Other; Difference in Percentage of Participants = -8.8, 95% CI [-16 to -1.9]
Statistical Analysis 2: Comparison: Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) vs Epoetin Alfa:Once Every Two Weeks (Q2W); Test type: Superiority or Other; Difference in Percentage of Participants = -10.0, 95% CI [-18.0 to -3.2]

ADVERSE EVENTS:
Time Frame: 44 weeks
Arm/Group | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) | Epoetin Alfa:Once Weekly (QW) | Epoetin Alfa:Once Every Two Weeks (Q2W)
Serious Adverse Events (participants affected / at risk) | 36/123 | 41/125 | 42/125
Other Adverse Events (participants affected / at risk) | 93/123 | 85/125 | 102/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) (N=123) | Epoetin Alfa:Once Weekly (QW) (N=125) | Epoetin Alfa:Once Every Two Weeks (Q2W) (N=125)
Cardiac failure congestive (Cardiac disorders) | 4 | 4 | 6
Myocardial Infarction (Cardiac disorders) | 0 | 2 | 5
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Subendocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 0 | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 4 | 3 | 5
Renal failure acute (Renal and urinary disorders) | 2 | 2 | 3
Obstructive uropathy (Renal and urinary disorders) | 1 | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 1
Convulsion (Nervous system disorders) | 1 | 1 | 0
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Encephalomalacia (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0
Arterial stenosis limb (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0
Vascular pseudoaneurysm ruptured (Vascular disorders) | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Device electrical finding (Injury, poisoning and procedural complications) | 0 | 0 | 1
Failure to capture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer metastitic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 1
Necrosis (General disorders) | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1 | 0
Walking disability (Social circumstances) | 1 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epoetin Alfa:Three Injections Weekly (TIW)/Once Weekly (QW) (N=123) | Epoetin Alfa:Once Weekly (QW) (N=125) | Epoetin Alfa:Once Every Two Weeks (Q2W) (N=125)
Urinary tract infection (Infections and infestations) | 9 | 15 | 14
Nasopharyngitis (Infections and infestations) | 4 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 13 | 13 | 10
Nausea (Gastrointestinal disorders) | 13 | 9 | 9
Vomiting (Gastrointestinal disorders) | 8 | 8 | 10
Constipation (Gastrointestinal disorders) | 8 | 3 | 14
Fatigue (General disorders) | 13 | 9 | 12
Oedema (General disorders) | 13 | 11 | 10
Oedema peripheral (General disorders) | 15 | 7 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 10 | 14
Metabolic acidosis (Metabolism and nutrition disorders) | 6 | 4 | 4
Dizziness (Nervous system disorders) | 12 | 7 | 16
Headache (Nervous system disorders) | 15 | 9 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 1 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6 | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 5
Hypertension (Vascular disorders) | 15 | 18 | 10
Hypotension (Vascular disorders) | 6 | 5 | 10
Insomnia (Psychiatric disorders) | 3 | 8 | 4
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions on the PI are pre- review of publications prior to public release. Sponsor can embargo trial result publication for up to 120 days. The PI may not publish the sponsor's confidential information without consent. In multi-center trials, individual PI's may publish results only if the study group has not published results 12 months after study completion, abandonment, or termination. The sponsor cannot require changes to the scientific content and cannot extend the embargo.